CLINICAL TRIAL: NCT01485497
Title: Evaluation of Obstructive Sleep Apnea With Long Range 3D Endoscopic Fourier Domain Optical Coherence Tomography (FDOCT)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: University of California, Irvine (Other)
Collaborators: VA Long Beach Healthcare System (U.S. Federal Agency); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Jun Zhang, PhD, Assistant Project Scientist, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20118075
Record Dates: First submitted 2011-08-02; First posted 2011-12-05 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Sleep Apnea
Keywords: APNEA
MeSH Terms: conditions — Sleep Apnea Syndromes; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3D endoscopic Fourier Domain OCT (Other): 3D endoscopic Fourier Domain OCT
  Interventions: Device: 3D endoscopic Fourier Domain OCT

INTERVENTIONS:
Device: 3D endoscopic Fourier Domain OCT — Evaluation of Obstructive Sleep Apnea

SUMMARY:
The purpose of this study is to determine whether the Optical coherence tomography (OCT) can image the structure and geometry of hollow organs of the upper airway in sleep disorder. The research can identify the obstruction sites that help the select the appropriate treatment for potential surgical candidates.

DETAILED DESCRIPTION:
The National Commission on Sleep Disorders Research estimated that 18 million Americans suffer from obstructive sleep apnea (OSA) The majority of them are undiagnosed and untreated at this time.

The current diagnostic gold standard for OSA is in-laboratory, a full night polysomnography (PSG). However, PSG is unable to provide information on upper airway structure and anatomy, and cannot identify the obstruction sites. OSA can lead to severe health complications including hypertension, heart failure, memory impairment, motor vehicle and work accidents, decreased work productivity, and increased risk of death.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female age 18-65 years has no history of obstructive sleep apnea
2. Male or Female age 18-65 years has been diagnose of mild to moderate obstructive sleep apnea
3. Male or Female age 18-65 years has been diagnose severe obstructive sleep apnea

Exclusion Criteria:

1. Pregnant women.
2. Breastfeeding women.
3. Unable to understand or give consent to the study.
4. Currently taking drugs that are sensitive to light.
5. Currently taking routine anti-convulsion, sedative or antihistamine drugs.
6. Currently taking immuno-suppressive drug therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
obstructive upper airways in sleep disordered | 8 hours
  The OCT can provide information on upper airway structure and anatomy, and identify the obstruction sites.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Principal Investigator — UCI Beckman Laser Institute